CLINICAL TRIAL: NCT00503516
Title: Multicenter, Double Blind, Randomized, Clinical Trial, Controlled With Placebo, to Evaluate the Effect of the Treatment With 320 mg/Day of Megestrol Acetate During 24 Weeks in the Weight Loss in Mixed Dementia Patients.
Brief Title: Study to Evaluate the Effect of Megestrol Acetate in Weight Loss in Dementia Patients
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Difficulties to recruit the patients following the inclusion criteria
Sponsor: Rottapharm Spain (Industry)
Responsible Party: Anna Anguera, Research Manager, Madaus, S.A.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BO-EC-DEM-02; EudraCT number:2006-005759-13
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Dementia
Keywords: weight loss, appetite, dementia, megestrol acetate
MeSH Terms: conditions — Dementia; Weight Loss | interventions — Megestrol Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Megestrol acetate 160 mg b.i.d. during 24 weeks
  Interventions: Drug: Megestrol acetate
- 2 (Placebo Comparator): 1 sachet of powder of placebo b.i.d. during 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Megestrol acetate — 1 sachet of powder containing 160 mg of megestrol acetate b.i.d. during 24 weeks
  Arms: 1
Drug: Placebo — 1 sachet of 160 mg of placebo b.i.d.
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the efficacy of megestrol acetate in the gain of body weight in patients with primary or mixed Dementia with a weight loss.

DETAILED DESCRIPTION:
In all geriatric patients with dementia it was prove a weight loss independently if they are institutionalized or not.There are some previous studies that indicates the effect of the megestrol acetate in the weight gain of patients with cachexia-anorexia related with neoplasia. It seems that the mechanism of development could be the same between these patients and patients with dementia. It was described an important role of a group of cytokines ( Il-6, leptin, neuropeptide Y, TNFalfa) in the development of this nutritional alteration.

Some previous pilots studies indicates that megestrol acetate has and effect in geriatric and dementia patients with a weight loss of at least 5% in the last 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed of primary or mixed dementia (CIE 10criteria)
* Weihgt loss >5% of habitual weight in the last 6 months and proteic-caloric malnutrition (MNA <17)
* Outpatients
* Patients that accept the participation in the study

Exclusion Criteria:

* Vascular pure Dementia and secondary dementias( vascular dementia, Parkinson disease,etc)
* Dementia in a terminal phase: category of FAST 7c in the Reisber scale
* Concomitant treatment with steroids, androgens or other drugs with progestagens
* Weight loss secondary to neoplasia

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the change in the body weight | 24 weeks

SECONDARY OUTCOMES:
To evaluate the change in the appetite | 24 weeks
To evaluate the change in biochemical markers: Il-6, Il-1, leptin, TNFalfa, neuropeptide Y, albumin and prealbumin | 24 weeks
Evaluate the change in the nutritional status (Mini-Nutritional Assessment) | 24 weeks
To evaluate the change in cognitive state ( Mini-Mental State Examination) | 24 weeks
To evaluate the safety of the treatment | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pau Sánchez, MD, Study Chair — Hospital Socio Sanitario del Hospitalet (Barcelona); Salvador Altimir, MD, Principal Investigator — Hospital Universitari Germans Trias i Pujol (Badalona); Ramón Cristófol, MD, Principal Investigator — Antic Hospital Sant Jaume i Santa Magdalena (Mataró); Olga Sabartés, MD, Principal Investigator — Hospital del Mar; Enrique Arriola, MD, Principal Investigator — Fundación Matia (San Sebastián); José Luis González, MD, Principal Investigator — Hospital Nuestra Señora de la Montaña (Cáceres); Esher Martínez, MD, Principal Investigator — Hospital de la Santa Creu (Tortosa); Roberto Petidier, MD, Principal Investigator — Hospital Universitario de Getafe (Madrid); Esperanza Martin, MD, Principal Investigator — Hospital Virgen del Valle (Toledo); Almudena Garnica, MD, Principal Investigator — Hospital Universitari San Joan de Reus (Tarragona); Regina Feijoo, MD, Principal Investigator — Hosp. Sta. Caterina Gerona; Anna Tantiña, MD, Principal Investigator — CAP Centelles (Barcelona)
Locations (1):
- Hospital Socio Sanitario del Hospitalet, El Hospitalet, Barcelona, Spain